CLINICAL TRIAL: NCT03568123
Title: A Prospective Randomized Control Study on CR vs MC Polyethylene Bearing With Persona Total Knee System in Total Knee Arthroplasty
Brief Title: A Comparison of the Persona Total Knee Arthroplasty System Using CR or MC Polyethylene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anders Troelsen (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor-Investigator, Anders Troelsen, Professor, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-16034695
Record Dates: First submitted 2018-05-17; First posted 2018-06-26 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: This project is carried out as a 2-arm randomized controlled single-blinded trial, in which the clinical and radiological outcomes after treatment of hip osteoarthritis with insertion of either 1) Persona Total Knee System with MC polyethylene bearing or 2) Persona Total Knee System with CR polyethylene bearing. Allocation of the participants to one of the two treatment groups is done intraoperatively. A computer-generated random allocation sequence will be used. Non-transparent envelopes are used for the randomization process.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are unaware of which prosthesis they receive and the research coordinator handling the collected questionnaires postoperatively is also unaware of which prosthesis the participant has received. The research assistant handling both standard RSA as well as dynamic RSA analysis is also unaware of which prosthesis the participant has received
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MC polyethylene bearing (Experimental): Persona Total Knee System with MC polyethylene bearing
  Interventions: Device: MC polyethylene bearing
- CR polyethylene bearing (Active Comparator): Persona Total Knee System with a CR polyethylene liner.
  Interventions: Device: CR polyethylene bearing

INTERVENTIONS:
Device: MC polyethylene bearing — Zimmer Biomet Persona Total Knee System with MC polyethylene bearing. Femoral component: Only cemented femoral components will be used for this study. Both standard as well as narrow femoral components will be used, depending on the patient anatomy.
  Tibial component: Only cemented tibial components will be used for this study. Polyethylene materials: Conventional polyethylene will be used for patients >65 years old and Vitamine-E infused poly insert for patients ≤ 65 years old.
  Arms: MC polyethylene bearing
Device: CR polyethylene bearing — Zimmer Biomet Persona Total Knee System with CR polyethylene bearing. Femoral component: Only cemented femoral components will be used for this study. Both standard as well as narrow femoral components will be used, depending on the patient anatomy.
  Tibial component: Only cemented tibial components will be used for this study. Polyethylene materials: Conventional polyethylene will be used for patients >65 years old and Vitamine-E infused poly insert for patients ≤ 65 years old.
  Arms: CR polyethylene bearing

SUMMARY:
Knee replacement is an established treatment for late stage osteoarthritis (OA) of the knee (Charnley et al. 1961). Recently, Zimmer-Biomet have introduced Persona Total Knee system with design changes that include asymmetric tibia plate, increased medial pivoting and more extensive choices in respect to poly thickness, all with the purpose to improve balancing, stability and longevity. One design change that is introduced is the medial congruent (MC) polyethylene to be used instead of standard cruciate retaining (CR) design. The theoretic proposed benefit of MC polyethylene bearing is improved kinematics mimicking native knee motion. However, currently no studies exist evaluating outcome following use of MC polyethylene bearing. Therefore such design changes and proposed benefits need to be evaluated in a prospective clinical trail, with focus on patient safety, satisfaction and implant durability.

In this project the investigators wish to:

Evaluate stability and fixation, intra-operative and postop complications, survivorship and patient reported outcome measures following primary total knee replacement using MC polyethylene bearing compared to CR polyethylene bearing with Persona Total Knee for treatment of knee osteoarthritis.

This project is carried out as a 2-arm randomized controlled single-blinded trial, in which the clinical and radiological outcomes after treatment of knee osteoarthritis with insertion of either 1) Persona Total Knee System with MC polyethylene bearing or 2) Persona Total Knee System with CR polyethylene bearing are compared. Recruitment of participants to this project is expected to begin in October 2016 or as soon as permission from the Regional Ethics Committee and the Danish Data Protections Agency is obtained. A total of 60 participants are to be included at Hvidovre University Hospital. Recruitment is expected completed after a period of 1.5 year. The project is expected to be completed 2 years after recruitment of the last participant (2019).

Participants are seen on an outpatient basis at 3 months, 1 and 2 years postoperatively. RSA is performed postoperatively and at all outpatient follow-ups. Dynamic RSA is performed at 1 year follow-up. The patients will be followed for survival through The Danish Knee Arthroplasty Registry.

This project is financed by Zimmer-Biomet®, Warsaw, Indiana, USA. The primary investigator of this project has independently initiated the project.

DETAILED DESCRIPTION:
Background Knee replacement is an established treatment for late stage osteoarthritis (OA) of the knee (Charnley et al. 1961). There are different approaches to prosthetic replacement and current practices and designs are often based on limited evidence (Plate et al. 2012). There have been individual cohort studies, indirect comparisons and retrospective studies to test the efficacy of a variety of different total knee replacement devices but there are very few high quality investigations of new paradigms or significant design change. Those studies that do exist have usually been undertaken to address a combination of design changes and many involve only short-term assessments (Mäkelä et al. 2008). Ongoing research and development programs for knee replacement are increasingly taking account of the needs of the changing characteristics of the late stage OA knee population.

There is an increasing demand for joint replacement in a younger population (Mäkelä et al. 2014). Due to the changing demographics of joint replacement, the population of younger patients are seeking options that not only correct their disease or deformity, but do not limit them in activity (Geerdink et al. 2009). Activities of daily living take higher priority in this patient group, and patients needing total joint replacement do not have many options that accommodate higher levels of activity.

Studies have shown that modern implant designs can potentially improve outcome. Therefore new implants are introduced to the marked with the theoretical benefit of improved implant survival and superior patient reported outcomes. Within Total knee arthroplasty, design changes are introduced in attempt to improve knee kinematics, improve alignment and functionality, but those potential improvements need to be evaluated Recently, Zimmer-Biomet have introduced Persona Total Knee system with design changes that include asymmetric tibia plate, increased medial pivoting and more extensive choices in respect to poly thickness, all with the purpose to improve balancing, stability and longevity. One design change that is introduced is the medial congruent (MC) polyethylene to be used instead of standard cruciate retaining (CR) design. The theoretic proposed benefit of MC polyethylene bearing is improved kinematics mimicking native knee motion. However, currently no studies exist evaluating outcome following use of MC polyethylene bearing. Therefore such design changes and proposed benefits need to be evaluated in a prospective clinical trail, with focus on patient safety, satisfaction and implant durability.

The purpose of the proposed Randomized Clinical Trial (RCT) is to evaluate the outcome and safety of a newly designed polyethylene bearing by comparing it with a control group of patients implanted with an established polyethylene bearing.

Device description

The devices to be used in this project are:

The Zimmer-Biomet Persona Total Knee System

The Zimmer-Biomet Persona Total Knee System is a novel total knee system developed by Zimmer-Biomet. Components are available in numerous designs for both systems, with cemented as well as cementless fixations and with numerous polyethylene inserts to accommodate the surgical demand based on patient characteristics. Both MC polyethylene bearing and CR polyethylene bearing will be used in this study.

Femoral component:

Only cemented femoral components will be used for this study. Both standard as well as narrow femoral components will be used, depending on the patient anatomy.

Tibial component:

Only cemented tibial components will be used for this study.

Polyethylene materials:

Conventional polyethylene will be used for patients >65 years old and Vitamine-E infused poly insert for patients ≤ 65 years old.

All devises are European Conformity (CE) marked and used as intended by the manufacturer.

Project design Project type This project is carried out as a 2-arm randomized controlled single-blinded trial, in which the clinical and radiological outcomes after treatment of hip osteoarthritis with insertion of either 1) Persona Total Knee System with MC polyethylene bearing or 2) Persona Total Knee System with CR polyethylene bearing. Allocation of the participants to one of the two treatment groups is done intraoperatively. Non-transparent envelopes are used for the randomization process. Participants are unaware of which prosthesis they receive and the research coordinator handling the collected questionnaires postoperatively is also unaware of which prosthesis the participant has received. The research assistant handling both standard RSA as well as dynamic RSA analysis is also unaware of which prosthesis the participant has received

Standard treatment Patients who decline to participate in the study as well as patients who are not included or excluded from the study will be treated with a standard Total Knee Arthroplasty (TKA) implant and standard surgical care. Persona Total Knee System with a CR polyethylene liner has been used as a standard implant of choice at Hvidovre Hospital since January 2016 for patients suited for a CR implant. Patients with insufficient posterior cruciate ligament (PCL) and other patients unsuited for a CR implant receive a posterior stabilized (LPS) NexGen TKA. All knees are performed in a standardized fast-track setup with the same surgical technique as described below, immediate mobilization after surgery and clinical and radiological controls after 3 months, 1 and 2 years.

Time schedule Recruitment of participants to this project is expected to begin in October 2016 or as soon as permission from the Regional Ethics Committee and the Danish Data Protections Agency is obtained. A total of 60 participants are to be included at Hvidovre University Hospital. Recruitment is expected completed after a period of 1 year. The project is expected to be completed 2 years after recruitment of the last participant (2019).

Participant termination It is recognized that the subject's participation in this study is entirely voluntary, and that she/he may refuse to participate and may withdraw from participation at any time without jeopardy to any future medical care. It is also recognized that the investigator, at his/her discretion, may withdraw a subject from this study based upon his/her professional judgment, e.g. in the event of deep infection leading to replacement of the prosthesis or long-term immobilization because of comorbidity. If a participant is withdrawn or rescinds their consent, a "Lost to Follow-up" case report form will be completed detailing the reason for the participant's withdrawal.

Data recording Data relevant for this project will be registered in a data sheet. An individual data sheet will be kept for each recruited participant. Data will also be aggregated and stored electronically. The storage of data will be done according to the rules posted by the Danish Data Protection Agency. This project will be notified to and approved by the Danish Data Protection Agency before recruitment of participants is initiated.

Participant population in Denmark Study population will consist of 60 participants with knee osteoarthritis set to receive primary total knee arthroplasty. The participants will be included at Hvidovre University Hospital, (see participating centers).

Number of participants Patients at are randomized to receive either 1) Persona Total Knee System with MC polyethylene bearing or 2) Persona Total Knee System with CR polyethylene bearing. Participants may be excluded intraoperatively if the PCL is found insufficient and LPS prosthesis is required.

In this 2-arm randomized controlled study the primary endpoint is implant migration measured by RSA. Secondary outcomes are: Oxford Knee Score (OKS), Oxford Knee Score -Activity & Participation Questionnaire (APQ), anchoring questions, EQ-5D, Forgotten Joint Score and knee motion measured using dynamic RSA.

The study's primary outcome measure is implant migration measured by RSA. If the minimally relevant total migration of the prosthesis measured by RSA is set to 0.2 mm then a total of 18 participants must be enrolled in each study group to show a statistically significant difference (95 % confidence, 80 % power). In this study 2 x 30 participants are included. This will insure sufficient statistical power despite intraoperative exclusion and dropout of 40% at last follow-up and .

The power calculation is based on reaching sufficient power when a comparison of the two study groups is carried out.

Participant inclusion All participants will receive oral and written information about the project before consent. It is the responsibility of the primary investigator that the information to the participant is adequate. Participants are included when signed consent from the participant is obtained. Project information is then given in an undisturbed environment (in a closed examination room) by an authorized investigator of this project. Project information is given at the first outpatient consultation, when treatment with insertion of a TKA is decided. A nurse is present when the information is given. Participants are informed about the right to having a dependent present when project information is given. Participants are informed that a period of consideration of at least 2 weeks is an opportunity along with the right to a second consultation. Signed consent, however, is to be given latest at admittance before surgery.

The oral information is in accordance with the written information and is adjusted to the age, educational level and social conditions of the participant. It is ensured that the participant has understood the content of both the oral and written information before signed consent is given.

It is recognized that the subject's participation in this study is entirely voluntary, and that she/he may refuse to participate and may withdraw from participation at any time without jeopardy to any future medical care. It is also recognized that the investigator, at his/her discretion, may withdraw a subject from this study based upon his/her professional judgment, e.g. in the event of deep infection leading to replacement of the prosthesis or long-term immobilization because of comorbidity. If a participant is withdrawn or rescinds their consent, a "Lost to Follow-up" case report form will be completed detailing the reason for the participant's withdrawal.

Data recordings Participants in this project are identified with an assigned allocation number. At the end of the project all patient related data are destroyed.

All sensitive personal data regarding participants will be stored in accordance with guidelines presented by the Personal Data Act. Personal data regarding participants will be treated anonymously. The project will be reported to the Danish Data Protection Agency. The primary investigator will process all data. Participants will receive oral and written information concerning the handling of sensitive personal data.

Statistics A professional statistical software package will be used when processing data in this project. Comparative statistics will be used based on the distribution of data.

Publications The results of this project are expected published in an international medical journal. The results of this project are also expected presented at national and international orthopedic conventions. If publication is not achieved, the results of this project (positive, negative or inconclusive) will be presented on the homepage of the investigator's institution.

Co-authorship is awarded according to the Vancouver rules.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological osteoarthritis of the knee set to receive a primary unilateral total knee replacement
* >18 years of age
* Participants must be able to speak and understand Danish
* Participants must be able to give informed consent and be cognitively intact
* Participants must be able to complete all post-operative controls
* Participants must not have severe comorbidities, American Society of Anesthesiologists Physical Status Classification System (ASA) score ≤ 3
* Clinically suitable to receive a Cruciate Retaining (CR) implant (no severe deformity and/or ligament instability)

Exclusion Criteria:

* Age under 18 years.
* Terminal illness
* Revision knee replacement surgery
* Rheumatoid Arthritis
* Traumatic etiology
* Prior surgery on the affected knee that includes osteosynthesis, anterior cruciate ligament (ACL) and/or posterior cruciate ligament (PCL) and/or collateral ligament surgery. Arthroscopy with meniscectomy / cartilage surgery / house cleaning is allowed.
* Altered pain perception and / or neurologic affection due to diabetes or other disorders.
* Patients will be excluded intraoperative if CR implant is not suitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Radiostereometric analysis (RSA) | 2 years after postoperatively
  Radiologically verified stability and fixation is measured as the Maximum total point motion (MTPM) using RSA

SECONDARY OUTCOMES:
Radiostereometric analysis (RSA) | 3 months postoperatively
  Radiologically verified stability and fixation is measured as the Maximum total point motion (MTPM) using RSA
Radiostereometric analysis (RSA) | 1 year postoperatively
  Radiologically verified stability and fixation is measured as the Maximum total point motion (MTPM) using RSA
Oxford Knee Score (OKS) | Change from preoperative to 3 months postoperative OKS
  The Oxford Knee Score (OKS) measures knee pain and function. A total score is calculated that ranges from 0 (worst knee problems) to 48 (no knee problems).
Oxford Knee Score (OKS) | Change from preoperative to 1 year postoperative OKS
  The Oxford Knee Score (OKS) measures knee pain and function. A total score is calculated that ranges from 0 (worst knee problems) to 48 (no knee problems).
Oxford Knee Score (OKS) | Change from preoperative to 2 years postoperative OKS
  The Oxford Knee Score (OKS) measures knee pain and function. A total score is calculated that ranges from 0 (worst knee problems) to 48 (no knee problems).
Oxford Knee Score - Activity & Participation Questionnaire (OKS-APQ) | Change from preoperative to 3 months postoperatively
  An add-on to the Oxford Knee Score will evaluate the patients activity and participation restrictions due to their knee problem. A total score ranging from 0 (worst) to 100 (best) is calculated.
Oxford Knee Score - Activity & Participation Questionnaire (OKS-APQ) | Change from preoperative to 1 year postoperatively
  An add-on to the Oxford Knee Score will evaluate the patients activity and participation restrictions due to their knee problem. A total score ranging from 0 (worst) to 100 (best) is calculated.
Oxford Knee Score - Activity & Participation Questionnaire (OKS-APQ) | Change from preoperative to 2 years postoperatively
  An add-on to the Oxford Knee Score will evaluate the patients activity and participation restrictions due to their knee problem. A total score ranging from 0 (worst) to 100 (best) is calculated.
EuroQol 5-dimension (EQ-5D) | Change from preoperative to 3 months postoperatively
  The EuroQol 5-dimension (EQ-5D) is a generic questionnaire that measures the overall health-related quality of life. A total score is calculated ranging from -0.624 (worst) to 1 (best).
EuroQol 5-dimension (EQ-5D) | Change from preoperative to 1 year postoperatively
  The EuroQol 5-dimension (EQ-5D) is a generic questionnaire that measures the overall health-related quality of life. A total score is calculated ranging from -0.624 (worst) to 1 (best).
EuroQol 5-dimension (EQ-5D) | Change from preoperative to 2 years postoperatively
  The EuroQol 5-dimension (EQ-5D) is a generic questionnaire that measures the overall health-related quality of life. A total score is calculated ranging from -0.624 (worst) to 1 (best).
Forgotten Joint Score (FJS) | Change from preoperative to 3 months postoperatively
  The Forgotten Joint Score (FJS) measures the degree of joint awareness. A total score is calculated that ranges from 0 (high knee awareness) to 100 (low knee awareness).
Forgotten Joint Score (FJS) | Change from preoperative to 1 year postoperatively
  The Forgotten Joint Score (FJS) measures the degree of joint awareness. A total score is calculated that ranges from 0 (high knee awareness) to 100 (low knee awareness).
Forgotten Joint Score (FJS) | Change from preoperative to 2 year postoperatively
  The Forgotten Joint Score (FJS) measures the degree of joint awareness. A total score is calculated that ranges from 0 (high knee awareness) to 100 (low knee awareness).
Dynamic RSA | 1 year postoperatively
  Knee motion following primary total knee replacement in both treatment Groups will be measured using fluoroscopic dynamic RSA analysis.
Radiolucency / osteolysis | immediate postoperatively and 1 and 2 years postoperatively
  Radiographically verified radiolucency / osteolysis
Adverse Events | Through study completion, up to 2 years postoperatively
  Adverse Events including intraoperative complications and revisions at any post-operative time points.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Troelsen, Professor, Principal Investigator — Department of orthopaedic surgery; Kirill Gromov, PhD, Principal Investigator — Department of orthopaedic surgery
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charnley J. Arthroplasty of the hip. A new operation. Lancet. 1961 May 27;1(7187):1129-32. doi: 10.1016/s0140-6736(61)92063-3. No abstract available. PMID 15898154
- [Background] Plate JF, Seyler TM, Stroh DA, Issa K, Akbar M, Mont MA. Risk of dislocation using large- vs. small-diameter femoral heads in total hip arthroplasty. BMC Res Notes. 2012 Oct 5;5:553. doi: 10.1186/1756-0500-5-553. PMID 23039109
- [Background] Makela KT, Eskelinen A, Pulkkinen P, Paavolainen P, Remes V. Total hip arthroplasty for primary osteoarthritis in patients fifty-five years of age or older. An analysis of the Finnish arthroplasty registry. J Bone Joint Surg Am. 2008 Oct;90(10):2160-70. doi: 10.2106/JBJS.G.00870. PMID 18829914
- [Background] Geerdink CH, Grimm B, Vencken W, Heyligers IC, Tonino AJ. Cross-linked compared with historical polyethylene in THA: an 8-year clinical study. Clin Orthop Relat Res. 2009 Apr;467(4):979-84. doi: 10.1007/s11999-008-0628-2. Epub 2008 Nov 22. PMID 19030941
- [Background] Makela KT, Matilainen M, Pulkkinen P, Fenstad AM, Havelin L, Engesaeter L, Furnes O, Pedersen AB, Overgaard S, Karrholm J, Malchau H, Garellick G, Ranstam J, Eskelinen A. Failure rate of cemented and uncemented total hip replacements: register study of combined Nordic database of four nations. BMJ. 2014 Jan 13;348:f7592. doi: 10.1136/bmj.f7592. PMID 24418635